CLINICAL TRIAL: NCT02401529
Title: Effect of Steroids on Post-tonsillectomy Morbidities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Fahd General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Faris Bahammam, Dr, King Fahd General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Bahammam-1
Record Dates: First submitted 2015-03-21; First posted 2015-03-30 (Estimated); Results first posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting
Keywords: Dexamethasone; Prednisolone; Tonsillectomy Nausea; Pain, Postoperative; Postoperative Nausea and Vomiting; Randomized controlled trial; Post-tonsillectomy pain; delayed feeding
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Dexamethasone; Calcium Dobesilate; Prednisolone; Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV dexamethasone and oral Prednisolone (Experimental): Single dose of intravenous dexamethasone given immediately following surgery (0.15 mg/kg), followed by oral Prednisolone (0.25mg/kg/day for 7 days then tapering for next 7 days) and paracetamol (acetaminophen 15 mg/kg/dose every 6 hours).
  Interventions: Drug: IV dexamethasone; Drug: Oral prednisolone; Drug: Paracetamol
- Placebo (Active Comparator): Placebo (IV saline) and paracetamol (acetaminophen 15 mg/kg/dose every 6 hours).
  Interventions: Drug: Paracetamol; Drug: IV saline

INTERVENTIONS:
Drug: IV dexamethasone — 0.15 mg/kg
  Other Names: Decadron
  Arms: IV dexamethasone and oral Prednisolone
Drug: Oral prednisolone — 0.25mg/kg/day for 7 days then tapering for next 7 days
  Other Names: Predosone
  Arms: IV dexamethasone and oral Prednisolone
Drug: Paracetamol — acetaminophen 15 mg/kg/dose every 6 hours
  Other Names: Adol
Drug: IV saline — IV saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effect of postoperative systemic rapid onset and short acting dexamethasone followed by a tapering dose of oral prednisolone on post-tonsillectomy morbidities. Half of the patients who comply with the inclusion criteria were selected to receive a single postoperative dose of intravenous dexamethasone followed by oral steroids; the second group received placebo.

DETAILED DESCRIPTION:
The effect of preoperative systemic steroids on post-tonsillectomy morbidities such as pain, nausea, vomiting and delayed feeding was proven. However, this study aims to evaluate the effect of postoperative systemic rapid onset and short acting dexamethasone followed by a tapering dose of oral prednisolone on the aforementioned morbidities and on decreasing the duration and costs of hospital stays. patients who were in the waiting list for tonsillectomy procedure were screened for medical history and those who comply with the inclusion criteria were randomly assigned into two equal groups of 50 patients each. One group was selected to receive a single postoperative dose of intravenous dexamethasone followed by oral steroids; the second group received placebo. Questionnaires investigating postoperative pain, nausea, vomiting, and oral intake were answered by patients, parents or guardians where applicable.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the waiting list for tonsillectomy under general anesthesia who accepted to participate in the study.

Exclusion Criteria:

* Patients who are allergic to steroids or those who have medical conditions which contraindicate the use of steroid i.e diabetes mellitus, gastritis, or hypertension and those who were on exogenous steroid supplements.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Faris A Bahammam, MD, Principal Investigator — ORL and Head & Neck Surgeon

REFERENCES:
- [Background] Elhakim M, Ali NM, Rashed I, Riad MK, Refat M. Dexamethasone reduces postoperative vomiting and pain after pediatric tonsillectomy. Can J Anaesth. 2003 Apr;50(4):392-7. doi: 10.1007/BF03021038. English, French. PMID 12670818
- [Background] Weimert TA, Babyak JW, Richter HJ. Electrodissection tonsillectomy. Arch Otolaryngol Head Neck Surg. 1990 Feb;116(2):186-8. doi: 10.1001/archotol.1990.01870020062016. PMID 2297411
- [Background] Leach J, Manning S, Schaefer S. Comparison of two methods of tonsillectomy. Laryngoscope. 1993 Jun;103(6):619-22. doi: 10.1288/00005537-199306000-00008. PMID 8502095
- [Background] Jordan K, Sippel C, Schmoll HJ. Guidelines for antiemetic treatment of chemotherapy-induced nausea and vomiting: past, present, and future recommendations. Oncologist. 2007 Sep;12(9):1143-50. doi: 10.1634/theoncologist.12-9-1143. PMID 17914084
- [Background] Baxendale BR, Vater M, Lavery KM. Dexamethasone reduces pain and swelling following extraction of third molar teeth. Anaesthesia. 1993 Nov;48(11):961-4. doi: 10.1111/j.1365-2044.1993.tb07474.x. PMID 8250191
- [Background] Browning GG. Prophylactic steroids and/or antibiotics to reduce post-tonsillectomy morbidity: a yet unanswered conundrum. Clin Otolaryngol. 2010 Oct;35(5):417. doi: 10.1111/j.1749-4486.2010.02211.x. No abstract available. PMID 21108754
- [Background] Hermans V, De Pooter F, De Groote F, De Hert S, Van der Linden P. Effect of dexamethasone on nausea, vomiting, and pain in paediatric tonsillectomy. Br J Anaesth. 2012 Sep;109(3):427-31. doi: 10.1093/bja/aes249. PMID 22879656
- [Background] Park SK, Kim J, Kim JM, Yeon JY, Shim WS, Lee DW. Effects of oral prednisolone on recovery after tonsillectomy. Laryngoscope. 2015 Jan;125(1):111-7. doi: 10.1002/lary.24958. Epub 2014 Oct 7. PMID 25291409
- [Background] Andersen R, Krohg K. Pain as a major cause of postoperative nausea. Can Anaesth Soc J. 1976 Jul;23(4):366-9. doi: 10.1007/BF03005916. PMID 7347
- [Background] McKean S, Kochilas X, Kelleher R, Dockery M. Use of intravenous steroids at induction of anaesthesia for adult tonsillectomy to reduce post-operative nausea and vomiting and pain: a double-blind randomized controlled trial. Clin Otolaryngol. 2006 Feb;31(1):36-40. doi: 10.1111/j.1749-4486.2006.01141.x. PMID 16441800
- [Background] Beirne OR, Hollander B. The effect of methylprednisolone on pain, trismus, and swelling after removal of third molars. Oral Surg Oral Med Oral Pathol. 1986 Feb;61(2):134-8. doi: 10.1016/0030-4220(86)90173-8. PMID 3457335
- [Background] Campbell WI, Kendrick RW. Postoperative dental pain--a comparative study of anti-inflammatory and analgesic agents. Ulster Med J. 1991 Apr;60(1):39-43. PMID 1853495
- [Background] Henzi I, Walder B, Tramer MR. Dexamethasone for the prevention of postoperative nausea and vomiting: a quantitative systematic review. Anesth Analg. 2000 Jan;90(1):186-94. doi: 10.1097/00000539-200001000-00038. PMID 10625002
- [Background] Alexander TH, Weisman MH, Derebery JM, Espeland MA, Gantz BJ, Gulya AJ, Hammerschlag PE, Hannley M, Hughes GB, Moscicki R, Nelson RA, Niparko JK, Rauch SD, Telian SA, Brookhouser PE, Harris JP. Safety of high-dose corticosteroids for the treatment of autoimmune inner ear disease. Otol Neurotol. 2009 Jun;30(4):443-8. doi: 10.1097/MAO.0b013e3181a52773. PMID 19395984
- [Background] Thomas S, Beevi S. Epidural dexamethasone reduces postoperative pain and analgesic requirements. Can J Anaesth. 2006 Sep;53(9):899-905. doi: 10.1007/BF03022833. PMID 16960268
- [Background] Rich WM, Abdulhayoglu G, DiSaia PJ. Methylprednisolone as an antiemetic during cancer chemotherapy--a pilot study. Gynecol Oncol. 1980 Apr;9(2):193-8. doi: 10.1016/0090-8258(80)90027-x. No abstract available. PMID 7189499
- [Background] Fredrikson M, Hursti T, Furst CJ, Steineck G, Borjeson S, Wikblom M, Peterson C. Nausea in cancer chemotherapy is inversely related to urinary cortisol excretion. Br J Cancer. 1992 May;65(5):779-80. doi: 10.1038/bjc.1992.165. No abstract available. PMID 1586608
- [Background] Harris AL. Cytotoxic-therapy-induced vomiting is mediated via enkephalin pathways. Lancet. 1982 Mar 27;1(8274):714-6. doi: 10.1016/s0140-6736(82)92625-3. No abstract available. PMID 6122010
- [Background] Splinter W, Roberts DJ. Prophylaxis for vomiting by children after tonsillectomy: dexamethasone versus perphenazine. Anesth Analg. 1997 Sep;85(3):534-7. doi: 10.1097/00000539-199709000-00010. PMID 9296405
- [Background] Ahmad S, De Oliveira GS Jr, Fitzgerald PC, McCarthy RJ. The effect of intravenous dexamethasone and lidocaine on propofol-induced vascular pain: a randomized double-blinded placebo-controlled trial. Pain Res Treat. 2013;2013:734531. doi: 10.1155/2013/734531. Epub 2013 Jul 15. PMID 23956857
- [Background] Fazel MR, Yegane-Moghaddam A, Forghani Z, Aghadoost D, Mahdian M, Fakharian E. The effect of dexamethasone on postoperative vomiting and oral intake after adenotonsillectomy. Int J Pediatr Otorhinolaryngol. 2007 Aug;71(8):1235-8. doi: 10.1016/j.ijporl.2007.04.015. Epub 2007 Jun 1. PMID 17544156
- [Background] Hashmi MA, Ahmed A, Aslam S, Mubeen M. Post-tonsillectomy pain and vomiting:role of pre-operative steroids. J Coll Physicians Surg Pak. 2012 Aug;22(8):505-9. PMID 22868016
- [Background] Kaan MN, Odabasi O, Gezer E, Daldal A. The effect of preoperative dexamethasone on early oral intake, vomiting and pain after tonsillectomy. Int J Pediatr Otorhinolaryngol. 2006 Jan;70(1):73-9. doi: 10.1016/j.ijporl.2005.05.013. Epub 2005 Jun 24. PMID 15979735
- [Background] Steward DL, Welge JA, Myer CM. Steroids for improving recovery following tonsillectomy in children. Cochrane Database Syst Rev. 2003;(1):CD003997. doi: 10.1002/14651858.CD003997. PMID 12535500
- [Background] Scarlett M, Tennant I, Ehikhametalor K, Nelson M. Vomiting post tonsillectomy at the University Hospital of the West Indies. West Indian Med J. 2005 Jan;54(1):59-64. doi: 10.1590/s0043-31442005000100012. PMID 15892392

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 116 participants were initially considered for the study. However, only 100 were considered in the final results. some were excluded due to not matching inclusion criteria. others failed to attend follow up visits, adhere to treatment protocol or complete the questionnaire as required.
  Please refer to section ( period 1) for further details.
Period: Overall Study
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Started | 59 | 57
Completed | 50 | 50
Not Completed | 9 | 7
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 6
Not completed — Protocol Violation | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Full Range); unit: years] | 8.5 [5 to 19] | 8.7 [5 to 17] | 8.6 [5 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 34 | 29 | 63

OUTCOME MEASURES:

1. Primary Outcome: Maximum Severity of Post-operative Pain
Description: 5 grades (pain free, low disability and low intensity, low disability and high intensity, high disability and moderate intensity, high disability and severly limiting)
Time Frame: The severest pain grade felt within a week
Measure: Number; unit: participants
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  Low disability and low intensity | 37 | 26
  high disability and moderate intensity | 13 | 21
  high disability and high intensity | 0 | 3
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.033, Chi-squared

2. Primary Outcome: Duration of Post-operative Pain
Description: 4 selections (1 day, 2 days, 3 days, if more specify)
Time Frame: number of days at which pain was experienced within the the 1st sevn days post -surgery
Measure: Number; unit: participants
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  one day | 36 | 23
  two days | 11 | 19
  three days | 3 | 8
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.026, Chi-squared

3. Primary Outcome: Occurence of Post-operative Nausea
Description: Postoperative nausea occurence (yes, no)
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  yes | 17 | 29
  no | 33 | 21
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.016, Chi-squared

4. Primary Outcome: Onset of Post-operative Nausea
Description: Postoperative nausea onset (no nausea, immediate, 1st day, 2nd day, 3rd day, 4th day, 5th day, 6th day, 7th day)
Time Frame: onset of 1st ocurence of nausea attack within the 1st week post-surgery
Measure: Number; unit: participants
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  no nausea | 33 | 21
  immediately | 10 | 8
  1st day | 4 | 11
  immediately and 1st day | 3 | 10
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.019, Chi-squared

5. Primary Outcome: Duration of Post-operative Nausea
Description: Postoperative nausea duration (no nausea,1 day, 2 days, 3 days, 4 days, if more specify)
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  no nausea | 33 | 21
  one day | 3 | 8
  two days | 14 | 15
  three days | 0 | 6
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.012, Chi-squared

6. Primary Outcome: Occurence of Postoperative Vomiting
Description: Postoperative vomiting occurrence (yes, no)
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  yes | 25 | 36
  no | 25 | 14
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.024, Chi-squared

7. Primary Outcome: Total Number of Post-operative Vomiting Episodes
Description: Postoperative vomiting number of attacks (no vomiting,1, 2, 3, if more specify)
Time Frame: total number of post-operative vomiting episodes which were experienced within the 1st week post-surgery
Measure: Number; unit: participants
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  no vomiting | 25 | 14
  once | 13 | 9
  twice | 7 | 19
  three times | 4 | 8
  more than 3 times | 1 | 0
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.02, Chi-squared

8. Secondary Outcome: Onset of 1st Post-operative Oral Intake
Description: feeding onset (1st day i. surgery day, 2nd day, 3rd day)
Time Frame: Onset of 1st post-operative oral intake recorded within the 1st 3days post-surgery
Measure: Number; unit: participants
Groups:
- IV Dexamethasone and Oral Prednisolone: Single dose of intravenous dexamethasone given immediately following surgery (0.15 mg/kg), followed by oral Prednisolone (0.25mg/kg/day for 7 days then tapering for next 7 days) and paracetamol (acetaminophen 15 mg/kg/dose every 6 hours).
  IV dexamethasone: 0.15 mg/kg
  Oral prednisolone: 0.25mg/kg/day for 7 days then tapering for next 7 days
  Paracetamol: acetaminophen 15 mg/kg/dose every 6 hours
  Number of participants when started 59
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  surgery day | 46 | 37
  1st day after surgery | 4 | 13
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.017, Chi-squared

9. Secondary Outcome: Average Amount of Meal Per Day
Description: adequacy of meals (inadequate, adequate)
Time Frame: 3 days
Measure: Number; unit: participants
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  inadequate | 16 | 27
  adequate | 34 | 23
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.026, Chi-squared

10. Secondary Outcome: Average Frequency of Meals Per Day
Description: average frequency of meals (1 meal, 2 meals, if more specify)
Time Frame: average number of meals consumed per day for the 1st three days post-surgery
Measure: Number; unit: participants
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Number analyzed (Participants) | 50 | 50
participants
  1 meal | 2 | 1
  2 meals | 20 | 34
  3 meals | 28 | 15
Statistical Analysis 1: Comparison: IV Dexamethasone and Oral Prednisolone vs Placebo; Test type: Superiority or Other; p = 0.019, Chi-squared

ADVERSE EVENTS:
Arm/Group | IV Dexamethasone and Oral Prednisolone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Dexamethasone and Oral Prednisolone (N=50) | Placebo (N=50)
Infection (Surgical and medical procedures) | 0 (0) | 0 (0)
Excess stomach acid (Gastrointestinal disorders) | 0 (0) | 0 (0)
Bleeding (Surgical and medical procedures) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes